CLINICAL TRIAL: NCT06379789
Title: A Two-Part Open-Label Study of REGV131-LNP1265, A CRISPR/Cas9 Based Coagulation Factor IX Gene Insertion Therapy in Participants With Hemophilia B
Brief Title: A Study to Investigate the Safety and Effectiveness of a Coagulation Factor IX Gene Insertion Therapy (REGV131-LNP1265) in Pediatric, Adolescent and Adult Participants With Hemophilia B
Acronym: BEYOND-9
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R131L1265-HEMB-2318; 2023-507260-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia B
Keywords: Severe and moderately severe congenital hemophilia B; FIX functional activity
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: Cohort 1 Dose Escalation for RDE (Experimental): Starting dose to determine the RDE of REGV131-LNP1265 and further assess the safety, tolerability, and FIX functional activity data at the RDE
  Interventions: Drug: REGV131; Drug: LNP1265
- Part 1: Cohort 2 Dose Escalation for RDE (Experimental): Dose 2 of ascending dose level cohorts to determine the RDE of REGV131-LNP1265 and further assess the safety, tolerability, and FIX functional activity data at the RDE
  Interventions: Drug: REGV131; Drug: LNP1265
- Part 1: Cohort 3 Dose Escalation for RDE (Experimental): Dose 3 of ascending dose level cohorts to determine the RDE of REGV131-LNP1265 and further assess the safety, tolerability, and FIX functional activity data at the RDE
  Interventions: Drug: REGV131; Drug: LNP1265
- Part 1: Cohort 4 Dose Escalation for RDE (Experimental): Dose 4 of ascending dose level cohorts to determine the RDE of REGV131-LNP1265 and further assess the safety, tolerability, and FIX functional activity data at the RDE
  Interventions: Drug: REGV131; Drug: LNP1265
- Part 2: Dose Expansion A (Experimental): Participants ≥18 Years of Age will receive the RDE of REGV131-LNP1265 determined by Part 1
  Interventions: Drug: REGV131; Drug: LNP1265
- Part 2: Dose Expansion B (Experimental): Participants ≥12 to <18 Years of Age will receive the administered weight-adjusted RDE of REGV131-LNP1265 determined by Part 1
  Interventions: Drug: REGV131; Drug: LNP1265
- Part 2: Dose Expansion C (Experimental): Participants ≥2 to <12 Years of Age will receive the administered weight-adjusted RDE of REGV131-LNP1265 determined by Part 1
  Interventions: Drug: REGV131; Drug: LNP1265

INTERVENTIONS:
Drug: REGV131 — Single dose administered via intravenous (IV) infusion before LNP1265
Drug: LNP1265 — Single dose administered via IV infusion following REGV131

SUMMARY:
Participants in this study have a genetic mutation, specifically in the coagulation (blood clotting) Factor 9 gene that causes severe or moderately severe hemophilia B. This study is researching an experimental gene insertion therapy (the adding of a gene into your DNA) called REGV131-LNP1265, also called the "study drug". Gene insertion therapy aims to teach the body how to produce clotting factor long-term, without the need for factor replacement therapy.

The main aim of this study is to find a safe and well-tolerated dose of the study drug by checking the side effects that may happen from taking it.

The study is looking at several other research questions including:

* How much study drug is in the blood at different times
* Whether the body makes antibodies against parts of the study drug, which could make the drug less effective or could lead to side effects. Antibodies are proteins produced by the body's immune system in response to a foreign substance
* Whether the body makes antibodies against the clotting factor replacement therapy
* How quality of life is affected by hemophilia B and if it changes after taking study drug
* How joint health is affected by hemophilia B and if it changes after taking study drug
* How often visits are required for the emergency room, urgent care center, physician's office, hospital, telephone or online are required as a result of bleeding events, and if the frequency changes after taking study drug
* How often factor replacement therapy is needed, both on a regular basis for prevention of bleeding, and as needed to treat bleeding events (and it if changes after taking study drug)
* Whether there is a difference in 2 different methods for measuring Factor 9 activity in the blood

DETAILED DESCRIPTION:
The study will be conducted with a 2-part adaptive design, with enrollment of patients into sequential parts of the study.

Part 1: Dose Escalation and Dose Confirmation in adult patients ≥18 years of age

* Dose Escalation Cohorts to determine the recommended dose for expansion (RDE) of REGV131-LNP1265
* Dose Confirmation Cohort to gain further confidence in safety, tolerability, and Coagulation Factor IX (FIX) functional activity data at the RDE

Part 2: Dose Expansion at the RDE

* Part 2A: Adult patients ≥18 years of age: RDE of REGV131-LNP1265, as determined in Part 1
* Part 2B: Adolescent patients <18 and ≥12 years of age will be administered weight-adjusted RDE
* Part 2C: Adolescent and Pediatric patients ≥2 to <12 years may be enrolled in an age staggered sequential manner; first participants aged ≥6 to <12 years and then participants ≥2 to <6 years of age and will receive a weight-adjusted RDE

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of severe or moderately severe hemophilia B with medical history of FIX functional activity (≤2% or <0.02 IU/mL) or documented genotype known to produce severe hemophilia B
2. Currently taking FIX prophylaxis and previous experience with FIX therapy, as defined in the protocol
3. Participation in the lead-in period of this interventional study OR a separate lead-in study (R0000-HEMB-2187 [NCT05568459]) for at least 6 months for ABR data while taking FIX prophylaxis, as defined in the protocol

Key Exclusion Criteria:

1. History of FIX inhibitor (clinical or laboratory-based assessment) on 2 or more occasions
2. Bethesda inhibitor titer greater than the upper limit of normal (ULN) at screening
3. Detectable pre-existing antibodies to the adeno-associated virus serotype 8 (AAV8) capsid; as measured by enzyme-linked immunosorbent assay (ELISA) at prescreening (or final lead-in visit, if applicable).
4. Any significant underlying liver disease such as: cholestatic liver disease, liver cirrhosis, portal hypertension, splenomegaly, hepatic encephalopathy
5. Evidence of advanced liver fibrosis, as defined in the protocol
6. Evidence of cirrhosis and/or portal hypertension as assessed by abdominal ultrasound at screening or measured within 6 months prior to the screening visit
7. History of arterial or venous thrombo-embolic events, as defined in the protocol
8. History of hypersensitivity to corticosteroids or known medical condition that requires chronic administration of corticosteroids
9. Previously received any AAV gene-based therapy or intends to receive approved or investigational AAV-based gene therapy other than REGV131-LNP1265 during the study period

NOTE: Other Inclusion/Exclusion Protocol Defined Criteria Apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male gender at birth:
  Part 1: > 18 years of age, irrespective of weight Part 2A: > 18 years of age, irrespective of weight Part 2B: ≥12 to <18 years of age with weight ≥45 kg Part 2C: ≥ 2 to < 12 years of age
Enrollment: 130 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2032-12-17 (Estimated); Study Completion 2032-12-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 104 Weeks
  Part 1, Part 2B and Part 2C
Severity of TEAEs | Up to 104 Weeks
  Part 1, Part 2B and Part 2C
Coagulation Factor IX (FIX) functional activity measured using the chromogenic substrate assay | At day 29
  Part 1
Change in FIX functional activity in plasma, measured using the chromogenic substrate assay | Baseline and at Week 26, after REGV131-LNP1265 dosing at the recommended dose for expansion (RDE)
  Part 2A, Part 2B and Part 2C
Annualized bleeding rate (ABR) following sustained FIX functional activity among participants receiving the RDE | Over 52 Weeks; Weeks 26 to 78 post-REGV131-LNP1265 dosing
  Part 2A, Part 2B and Part 2C

SECONDARY OUTCOMES:
Change in FIX functional activity in plasma measured using the chromogenic substrate assay | Baseline and at Week 26, after REGV131-LNP1265 dosing at the RDE
  Part 1
ABR following sustained FIX functional activity among participants receiving the RDE | Over 52 Weeks; Weeks 26 to 78 post-REGV131-LNP1265 dosing
  Part 1
FIX functional activity in plasma over time during the study period using the chromogenic substrate assay | Up to 104 Weeks
Annualized treated bleeding rate (tABR) following sustained FIX functional activity, among participants receiving the RDE | Over 52 Weeks; Weeks 26 to 78 post-REGV131-LNP1265 dosing
Annualized utilization (IU/kg/year) of FIX replacement therapy following sustained FIX functional activity among participants receiving the RDE | Over 52 Weeks; Weeks 26 to 78 post-REGV131-LNP1265 dosing
Remaining free of FIX replacement therapy among those receiving the RDE following sustained FIX expression | Over 52 Weeks; Weeks 26 to 78 post-REGV131-LNP1265 dosing
Remaining zero spontaneous bleeding events among those receiving the RDE over sustained FIX functional activity period | Over 52 Weeks; Weeks 26 to 78 post-REGV131-LNP1265 dosing
Concentrations of REGV131 components | Up to 29 Days
Concentrations of LNP1265 components | Up to 29 Days
Detection of antibodies to the F9 transgene product FIX protein | Up to 104 Weeks
Detection of total binding antibodies (TAbs) to the adeno-associated virus 8 (AAV8) capsid proteins | Up to 104 Weeks
Detection of neutralizing antibodies/transduction inhibitors (NAb/TI) to the adeno-associated virus 8 (AAV8) capsid proteins | Up to 104 Weeks
Detection of antibodies to LNP1265 | Up to 104 Weeks
Detection of antibodies to CRISPR-associated protein 9 (Cas9) protein | Up to 104 Weeks
Detection of vector DNA in blood | Up to 104 Weeks
  Part 1
Detection of vector DNA in saliva | Up to 104 Weeks
  Part 1
Detection of vector DNA in nasal secretions | Up to 104 Weeks
  Part 1
Detection of vector DNA in semen | Up to 104 Weeks
  Part 1
Detection of vector DNA in urine | Up to 104 Weeks
  Part 1
Detection of vector DNA in feces | Up to 104 Weeks
  Part 1
Incidence of TEAEs | Up to 104 Weeks
  Part 2A
Severity of TEAEs | Up to 104 Weeks
  Part 2A
Detection of vector DNA in relevant matrices based on data analysis of Part 1 Dose Confirmation Cohort | Up to 104 Weeks
  Part 2A
Detection of vector DNA in relevant matrices over time based on data analysis from adult cohorts over time | Up to 104 Weeks
  Part 2B and Part 2C

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (38):
- United States (13):
  - Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University California San Francisco, San Francisco, California
  - University of Colorado Hemophilia and Thrombosis Center, Aurora, Colorado
  - Yale HTC, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Tulane University School of Medicine, Louisiana Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
- Royal Prince Alfred Hospital, Haemophilia Treatment Centre, Camperdown, New South Wales, Australia
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - McGill University Health Center (MUHC), Montreal, Quebec
- France (2):
  - Hospices Civils de Lyon, Bron, Lyon
  - Hopital Necker, Paris, Île-de-France Region
- Germany (2):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - University Hospital Hamburg Eppendorf, Hamburg
- Italy (2):
  - Fondazione Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Ca Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Irccs Humanitas Research Hospital, Rozzano, Lombardy
- Spain (8):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Complejo Hospitalario Universitario de A Coruña (Edificio Teresa Herrera-Materno Infantil), A Coruña, Galicia
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Haemostasis and Thrombosis Unit, Hospital La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (7):
  - Glasgow Royal Infirmary - Clinical Research Facility, Glasgow, Scotland
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS FT, Cambridge
  - Pathology and Pharmacy Building, The Royal London Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - St. Thomas' Hospital, London
  - Hammersmith Hospital Comprehensive Care Centre, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Study Information Website — https://hemophilia-beyond-9.com/